CLINICAL TRIAL: NCT04603144
Title: Identification of Frailty Predictors of Adverse Health Outcomes in Community-dwelling Individuals Aged 50 and Over: the SUCCEED Prospective Cohort
Brief Title: Identification of Frailty Predictors of Adverse Health Outcomes in Community-dwelling Individuals Aged 50 and Over
Acronym: SUCCEED
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190906
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Community Dwelling Individuals Aged 50 and Over
Keywords: ageing; frailty; community dwelling; prevalence; prognosis
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction. Although ageing is a general phenomenon, a great inter individual variability on the quality of ageing can be observed. This substantial heterogeneity may be partly explained by extrinsic factors such as lifestyle, habits, physical activity, diet, which may play an important role in the age-associated declines. The concept of frailty was introduced to account for variability in the aging process. This clinical and biological syndrome reflects a decrease in the physiological reserve, and leads to an insidious, precarious equilibrium that can break down during a stressful life event. In older adults, frailty is known to be associated with an increased risk of adverse outcomes, such as falls, fractures, unplanned hospitalizations, and death. Several frailty domains may only be slightly altered, so that early-stage frailty is not necessarily clinically visible. The most commonly used operational definitions of frailty are based on two different conceptual frameworks. Fried's rules-based criteria correspond to a physical phenotype, whereas the "Rockwood accumulative model" defines frailty as the accumulation of multiple deficits. These tools were built for individuals aged 65 and over. However, frailty can also be found in younger adults. Although the early detection of frailty is potentially important (since the condition might be reversible in its early stages), frailty has not been extensively investigated among middle-aged individuals. Indeed, most of the literature studies have focused on older adults or on a small number of frailty parameters the investigators hypothesized that the factors determining the main ageing-related adverse events are already present in middle age.

The main objectives of the SUCCEED cohort are therefore to 1/investigate the prevalence of frailty parameters in community-dwelling individuals aged 50 and over, 2/ assess the parameters' prognostic value for future adverse health events, 3/ investigate frailty classifications in this population and assess the evolution of profiles over time Method. The SUCCEED survey is a French retrospective and prospective cohort that includes community-dwelling individuals aged 50 years or over consecutively attending an outpatient clinic ("successful ageing") in a geriatric teaching hospital in the Paris area, France. Baseline parameters are collected using a self-administered questionnaire followed by an interview, physical measurements, and performance tests conducted by trained nurses, and then a standardized clinical evaluation by a geriatrician. This clinical assessment includes evaluation of autonomy, cognition, mood, balance, mobility, muscle strength, nutrition, comorbidities, continence, sensory functions, bone density, sleeping disorders.

Patients who have attended the outpatient clinic from the 01/01/2010 to 14/01/2020 are retrospectively included in the cohort, the other ones are prospectively included.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 50 and over previously included in the SUCCEED survey as from 1/1/2010 and being followed up who do not refuse to allow their data to be used for research purposes
* subjects aged 50 and over coming for the first time to the successful ageing clinic who do not refuse to allow their data to be used for research purposes

Exclusion Criteria:

* Age below 50y
* Individuals who refuse to allow their data to be used for research purposes
* Legal guardianship
* Subjects not able to understand the study questionnaires, based on investigator's judgement
* Cognitive, mental or psychiatric condition that, based on investigator's judgement, would jeopardise study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community-dwelling individuals aged 50 years or over attending an outpatient clinic ("successful ageing") in a geriatric teaching hospital in the Paris area, France
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2035-09-30 (Estimated); Study Completion 2075-09-30 (Estimated)

PRIMARY OUTCOMES:
number of morbid events | from baseline,during 40 years of follow up maximum
  occurrence of 1 morbid event defined by the following composite criteria: death or institutionalization or pathological fracture (Pouteau-Colles type wrist, vertebral fracture or compression, femoral neck) or unscheduled hospitalization or non-accidental fall.

SECONDARY OUTCOMES:
Overall Survival | from baseline , during 40 years of follow up maximum
  occurence of Death

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - CHU HENRI MONDOR, Créteil, France